CLINICAL TRIAL: NCT00510081
Title: An Open Label Evaluation of the Safety and Efficacy of Calcium Hydroxylapatite (Radiesse®) Injection in the Correction of Jowl-Associated Chin Notches
Brief Title: An Evaluation of an Injectable Material for Correction of Wrinkles
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was not executed. No subjects were enrolled.
Sponsor: Northwestern University (Other)
Responsible Party: Murad Alam, MD, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1253-013
Record Dates: First submitted 2007-07-31; First posted 2007-08-01 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Jowls

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): subjects will receive filler injections
  Interventions: Device: Calcium Hydroxylapatite injection

INTERVENTIONS:
Device: Calcium Hydroxylapatite injection — filler injection
  Other Names: Radiesse

SUMMARY:
The objective of this study is to determine the effectiveness of a filler in improving wrinkles.

DETAILED DESCRIPTION:
The primary objective of this study is to determine whether focal injection of calcium hydroxylapatite (Radiesse®), an injectable biodegradable filler, into jowl-induced chin notches can result in safe, aesthetically pleasing, and long-lasting correction of these.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-65
* Have wrinkles
* The subjects are in good health.
* The subject has willingness and the ability to understand and provide informed consent for the use of their tissue and communicate with the investigator.

Exclusion Criteria:

* Subjects who have received within the past 3 months or are planning to receive in the next 6 months, botulinum toxin injections for correction of wrinkles.
* Subjects who have received within the past one year any soft tissue augmentation material into the chin and experimental area (defined as any area on the face below the lower lip vermilion, excluding the lateral lip marionette line up to 1 cm below this level).
* Subjects with prior history of nodule formation or hypersensitivity reactions to lidocaine or medium-term augmentation materials, including hyaluronic acid derivatives, poly-L-lactic acid, and calcium hydroxylapatite.
* Subjects who are currently using anticoagulation therapy.
* Subjects who have a history of bleeding disorders.
* Subjects who are unable to understand the protocol or to give informed consent.
* Subjects with mental illness.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-07; Primary Completion 2009-02; Study Completion 2009-02

PRIMARY OUTCOMES:
Correction of wrinkles | 1 week

SECONDARY OUTCOMES:
Development of adverse events | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University, Feinberg School of Medicine, Department of Dermatology